CLINICAL TRIAL: NCT04817371
Title: Analysis of Volatile Organic Compounds in Exhaled Air and Sweat: Interest in Rapid Screening for SARS-CoV-2 Infection.
Brief Title: Analysis of Volatile Organic Compounds in Exhaled Air and Sweat: Interest in Rapid Screening for COVID-19 Infection.
Acronym: VOCSARSCOVDep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021_0013
Record Dates: First submitted 2021-03-15; First posted 2021-03-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Symptomatic patients with positive PCR (Other): Patients with symptoms of COVID-19 and whose PCR result is positive
  Interventions: Device: Volatile Organic Compounds analysis (e-noses); Other: Canine odor detection of Volatile Organic Compounds; Device: Volatile Organic Compounds analysis (mass spectrometry); Device: Volatile Organic Compounds analysis in sweat (mass spectrometry)
- Symptomatic patients with positive PCR for other respiratory virus (Other): Patients with symptomatic respiratory disease of infectious origin with negative RT-PCR for SARS-CoV-2 and positive RT-PCR for other respiratory viruses
  Interventions: Device: Volatile Organic Compounds analysis (e-noses); Other: Canine odor detection of Volatile Organic Compounds; Device: Volatile Organic Compounds analysis (mass spectrometry); Device: Volatile Organic Compounds analysis in sweat (mass spectrometry)
- Asymptomatic patients or healthy volunteers (Other): Patients or healthy volunteers with negative RT-PCR and negative serology
  Interventions: Device: Volatile Organic Compounds analysis (e-noses); Other: Canine odor detection of Volatile Organic Compounds; Device: Volatile Organic Compounds analysis (mass spectrometry); Device: Volatile Organic Compounds analysis in sweat (mass spectrometry)
- Volunteers or patients vaccinated against COVID-19 (Other): Volunteers or patients vaccinated against COVID-19 (complete vaccination scheme)
  Interventions: Device: Volatile Organic Compounds analysis (e-noses); Other: Canine odor detection of Volatile Organic Compounds; Device: Volatile Organic Compounds analysis (mass spectrometry); Device: Volatile Organic Compounds analysis in sweat (mass spectrometry)

INTERVENTIONS:
Device: Volatile Organic Compounds analysis (e-noses) — VOC analysis in exhaled air with e-noses.
Other: Canine odor detection of Volatile Organic Compounds — VOC analysis in sweat by trained dogs.
Device: Volatile Organic Compounds analysis (mass spectrometry) — VOC analysis in exhaled air with mass spectrometry.
Device: Volatile Organic Compounds analysis in sweat (mass spectrometry) — VOC analysis in sweat with mass spectrometry.

SUMMARY:
In the context of the actual pandemia of the Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) which requires a better diagnostic strategy for the management of patients.

The study of volatile organic compounds (VOC) detected in exhaled air or in sweat, is an innovative research area for respiratory diseases. The analysis of VOC can be done either by the technique of the mass spectrometry which allows the identification of each VOC in the exhaled air or by the technique of electronic nose, simpler and faster, which provides an idea of the general profile of the VOC without identifying them. The VOC have shown their interest in some situations, such as diagnostic or prognostic tool in patients followed for thoracic tumorous pathology or bronchial or pulmonary vascular diseases.

Moreover, it has recently been shown that properly trained dogs would be able to detect an olfactory signature of SARS-CoV-2 infection with a specificity greater than 90%; this olfactory signature corresponds to VOCs detectable by the flair of dogs (Nosaïs-Covid19 study).

Validation of the diagnostic value of VOC analyzes by non-invasive and rapid methods (electronic nose analysis or mass spectrometry; detection by the scent of dogs) for the rapid detection and early diagnosis of a SARS-CoV-2 infection warrants the performance of this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Subject included in the Foch Hospital :
* Patients managed at the Foch Hospital with RT-PCR screening for SARS-CoV-2 infection
* Healthy volunteers among the hospital staff, asymptomatic, for whom an RT-PCR SARS-CoV-2 is indicated or recommended.
* Healthy hospital volunteers vaccinated against COVID (full vaccination schedule completed)
* At least 18 years of age;
* Fluency in the French language;
* Have signed a consent form;
* Be affiliated with a health insurance plan.

Exclusion Criteria:

* Pregnant woman
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The first co-objective of this experimental study is to determine if VOCs analyzed by electronic noses are of interest for the diagnosis of an infection by SARS-CoV-2 (COVID-19) infection. | 1 day
  Identification of VOC profiles specific to the SARS-CoV-2 (VOC analysis by electronic noses) on exhalates collected under resting breathing conditions between patients with symptoms suggestive of COVID-19 and SARS-CoV-2 infection confirmed by RT-PCR, those whose infection is ruled out on the basis of the negativity RT-PCR and clinical/radiological data (non-COVID control patients), and those with another symptomatic respiratory viral infection confirmed by positive PCR for viruses other than SARS-CoV-2 other than SARS-CoV-2.
The second co-objective of this experimental study is to determine if VOCs analyzed by mass spectrometry is of interest for the diagnosis of an infection by SARS-CoV-2 (COVID-19) infection. | 1 day
  Identification of VOC profiles specific to the SARS-CoV-2 (VOC analysis by mass spectrometry) on exhalates collected under resting breathing conditions between patients with symptoms suggestive of COVID and SARS-CoV-2 infection confirmed by RT-PCR, those whose infection is ruled out on the basis of the negativity RT-PCR and clinical/radiological data (non-COVID control patients), and those with another symptomatic respiratory viral infection confirmed by positive PCR for viruses other than SARS-CoV-2 other than SARS-CoV-2.

SECONDARY OUTCOMES:
Identify the nature of VOCs associated with infection by SARS-CoV-2 by mass spectrometry in exhaled air and in sweat | 1 day
  The equivalences and differences in nature of VOCs associated with infection with SARS-CoV-2 between exhaled air and sweat identified by mass spectrometry.
Assessment of the specificity and sensitivity of canine olfactory detection of COVs associated with infection by SARS-CoV-2 (COVID-19) | 1 day
  Success rate of dogs trained in detecting COVID-19 from sweat samples taken from participating patients.
  The status of patients (infected and uninfected with COVID-19 from the result of the PCR) will be compared to the result of the canine olfactory detection of COVID-19 in sweat samples.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Devillier, PhD, Principal Investigator — Hopital Foch
Locations (1):
- Foch hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: Undecided